CLINICAL TRIAL: NCT03969836
Title: Study of Regional Cerebral Oxygenation and Brain Blood Volume Changes During Cardiac Surgery Using the NeurOS System
Brief Title: Regional Cerebral Oxygenation and Brain Blood Volume During Cardiac Surgery Using the NeurOS System
Acronym: COBBV-CS
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Jiapeng Huang, Professor of Anesthesiology, University of Louisville
Other Study IDs: 19.0272
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Heart Diseases
Keywords: cardiac surgery cerebral oxygenation, brain blood volume; cerebral oxygenation; brain blood volume
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NeurOS Group: All patients will have both INVOS and NeurOS systems placed before and during cardiac surgery for monitoring cerebral oxygenation and brain blood volume.
  Interventions: Device: NeurOS system

INTERVENTIONS:
Device: NeurOS system — NeurOS system pads will be placed on patients' head for monitoring.

SUMMARY:
Study of Regional Cerebral Oxygenation and Brain Blood Volume changes during Cardiac Surgery using the NeurOS system

DETAILED DESCRIPTION:
1. Title of the Research Project： Study of regional Cerebral Oxygenation and Brain Blood Volume changes during Cardiac Surgery using the NeurOS system (COBBV-CS Trial)
2. Background/Problem Statement: The use of regional cerebral oxygenation (rSO2) monitoring has grown clinically, even becoming the standard of care in some institutions. Monitoring of intracranial tissue oxygenation is fundamentally possible because light in the near infrared spectrum (700-900nm) penetrates bone, muscle, and other tissue. Oxyhemoglobin and deoxyhemoglobin have distinct peak absorption spectra, but there is an isobestic wavelength (i.e., wavelength for which the peak absorption of light is similar for oxyhemoglobin and deoxyhemoglobin, approximately 810nm) for absorption by total hemoglobin. Determination of rScO2 thus is possible with transmission of just 2 wavelengths of near-infrared spectroscopy (NIRS) to determine the relative concentrations of oxyhemoglobin versus total hemoglobin. A decrease in rSO2 from baseline >20% or an absolute rSO2 value <50% often is reported in clinical investigation as representing a clinically meaningful reduction or "desaturation."

The data is controversial on the benefits of NIRS to prevent or reduce stroke or delirium after cardiac surgery. However, it must be realized the inherent limitations of monitors alone to impact clinical outcomes without a standardized intervention algorithm. Although multiple NIRS monitors are approved in the United States and other countries primarily for assessing the adequacy of cerebral oxygenation during surgery, their approval is not based on the indication of detecting and/or lowering the frequency of neurological complications. In regard to the latter, strokes are believed widely to result primarily from cerebral embolism and/or cerebral hypoperfusion. Importantly, both etiologies can contribute to cerebral injury in the same patient insofar as hypoperfusion may delay washout of microembolism and/or compromise collateral perfusion to the ischemic penumbra. Many strokes, though, occur in subcortical brain areas or at sites remote from the area of NIRS monitoring, and many occur in the postoperative period after NIRS monitoring has concluded.

In addition, technological advances with NIRS monitoring have continued and now include the ability to perform bedside cerebral autoregulation monitoring. Regional cerebral oxygenation provides a clinically acceptable surrogate of cerebral blood flow (CBF) for clinical autoregulation monitoring. Monitoring CBF autoregulation with rSO2 has many clinically attractive features, including the following: It is noninvasive, monitoring requires little caregiver intervention, and it has sufficient resolution to discriminate the lower autoregulatory threshold to prevent brain ischemia. On the other hand, simply raising mean blood pressure targets during CPB, however, may not necessarily be beneficial because for some individuals this may result in blood pressure above the upper limit of autoregulation, which potentially could lead to cerebral hyperperfusion, increasing cerebral embolic load and/or enhancing cerebral edema in the setting of systemic inflammatory response to cardiac surgery. Individualizing blood pressure during CPB based on physiological endpoints such as rSO2 monitoring, rather than empiric targets, may provide a means for modifying the risk for renal injury and major organ morbidity and possibly mortality.

Problem Statement: Disposable rSO2 sensors are costly and is becoming a rate limiting factor hindering its widespread clinical use. Reusable sensors like NeurOS cerebral oximetry are only a fraction of cost with similar performances in healthy volunteers. The investigators will use NeurOS in accordance with its approved labeling and indications by FDA. Cardiac surgery has significant variations and great clinical importance of cerebral oxygenation during different stages of surgery. Blood volume changes before, during and after cardiopulmonary bypass have not been studied previously and could provide critical information to prevent postoperative cognitive changes. The NeurOS system calculates the sum of attenuation of two wavelengths to provide brain blood volume index (BVI) continuously.

3. Objectives:

1. To compare the performance of NeurOS with INVOS system during cardiac surgery
2. To study the brain blood volume changes during cardiac surgery, which has never been studied before.

4. Study Design/Methodology: All cardiac surgical patients are already receiving INVOS cerebral oximetry monitoring during surgery at Jewish Hospital. Both INVOS and NeurOS pads will be placed on the same patient. Continuous monitoring of both cerebral oximetry data for the whole length of cardiac surgery will be recorded and saved in a USB drive for retrieval and analysis. Key point left and right-side cerebral oximetry data include: Baseline, Anesthesia Induction, Incision, Initiation cardiopulmonary bypass (CPB), Aortic Clamping, Coming off CPB and Skin Closure. These key points data will be extracted for comparison between NeurOS and INVOS in terms of percentage change from the baseline. In addition, a time-rSO2 graph will be plotted for each patient side by side with NeurOS and INVOS cerebral oxygenation for trend comparison.

1. . Sample selection and size: 100 consecutive cardiac surgical patients at Jewish Hospital, Louisville, KY (2 months to recruit)
2. . Describe the proposed intervention: Apply the single use NeurOS cerebral oximetry sensor adhesive onto patients' forehead who are going to have cardiac surgery in the operating room before anesthesia induction.
3. . Data collection procedures, instruments used, and methods for data quality control: Anesthesia providers (attending anesthesiologists, residents and CRNAs) provide routine anesthesia care for cardiac surgery. NeurOS and INVOS rSO2 reading are automatically recorded in the VO200-NeurOS Cerebral Oximetry Monitor and the INOVS Monitor respectively. Significant events (Baseline, Anesthesia Induction, Incision, Initiation cardiopulmonary bypass (CPB), Aortic Clamping, Coming off CPB and Skin Closure) will be marked manually by the anesthesia providers in individual systems. Brain blood volume index will be automatically recorded and retracted from the NeurOS system once surgery is over. All data will be downloaded from the system into an encrypted USB drive for storage and analysis. Data quality control will be ensured by the individual system alarms for poor signals and be corrected by anesthesia providers.
4. . Unit of analysis and observation: Cerebral Oxygenation in percentage of oxyhemoglobin. Brain blood volume index in the sum of attenuation of two wavelengths.

5. Subject Recruitment Methods: All patients presenting to Jewish Hospital for cardiac surgery will be contacted for potential recruitment on the day of surgery in the preoperative area.

6. Informed Consent Process/Complete Waiver Process: Informed consent will be provided to all participants.

7. Research Procedures:

In all consented patients, baseline cerebral oxygenation and brain blood volume index will be obtained at room air or baseline oxygen requirement level in NeurOS and INVOS systems. Both NeurOS and INVOS rSO2 and brain blood volume indexes will be continuously recorded and saved in the respective system throughout the whole cardiac surgery. General anesthesia will be induced by using O2 administered via face mask and IV fentanyl 1μg/ kg, propofol 2-3mg/kg and rocuronium 1mg/kg. Maintenance of anesthesia was achieved with inhaled isoflurane in air/oxygen mixture and muscle relaxation using intermittent boluses of rocuronium. Fentanyl will be used as supplemental analgesia. Normocapnic ventilation was maintained. Upon completion of surgery and weaning from cardio pulmonary bypass, titrated doses of protamine will be administered to reverse the anticoagulant action of heparin, targeting to achieve baseline preoperative Activated clotting Time.

After the surgery, all rSO2 and brain blood volume index data are downloaded into an encrypted USB drive for analysis and storage.

8. Minimizing Risks:

1. All HIPPA related information will be stored in a private computer in a password protected computer.
2. Cleaning of cables, monitors and reusable equipment are performed after each use.
3. Standard electrical precautions will be followed to prevent electrical shock to providers and patients.

9. Plan for Analysis of Results:

* Trend graphs of INVOS and NeurOS cerebral oximetry will be plotted together to compare whether they follow a similar trend. Cerebral oxygenation deviation from the baseline will be compared through statistical analysis to identify whether NeurOS performs as well as INVOS at these critical moments during cardiac surgery.
* Trend graphs of NeurOS brain blood volume, arterial blood pressure, central venous pressure and cerebral oxygenation will be plotted together to identify correlations among these parameters. Each key point brain blood volume index deviation from the baseline will be analyzed to identify whether above mentioned critical moments during cardiac surgery will affect the brain blood volume. Clinical outcomes data will be collected on 30-day mortality and strokes to identify whether the brain blood volume index directly affects clinical outcomes.
* Programs to be used for data analysis: Software R

  10. Research Materials, Records, and Privacy: Identify the sources of research material obtained from individually identifiable living human subjects: Prospective noninvasive data on cerebral oxygenation and brain blood volume during cardiac surgery. Please see data collection form.

Indicate what information (records, data, etc.) will be recorded and whether use will be made of existing records or data: Cerebral oxygenation and brain blood volume. They will be recorded in the medical charts.

Explain why this information is needed to conduct the study: These data are necessary to identify outcomes for these patients.

Specify how the data will be de-identified (if applicable), who has access to the data, where the data will be stored and how the researcher will protect both the data with respect to privacy and confidentiality. Address physical security measures (e.g., locked facility, limited access); data security (e.g., password-protection, data encryption); safeguards to protect identifiable research information (e.g., coding or links): Once required information is collected, HIPPA information will be deleted. All HIPPA related information will be stored in a private computer in a password protected computer. No links will be provided to the public.

11. References

1. Lewis C, Parulkar SD, Bebawy J, Sherwani S, Hogue CW. Cerebral Neuromonitoring During Cardiac Surgery: A Critical Appraisal With an Emphasis on Near-Infrared Spectroscopy. Journal of Cardiothoracic and Vascular Anesthesia. 2018;32:2313-2322

ELIGIBILITY:
Inclusion Criteria:

* Having cardiac surgery at Jewish Hospital, Louisville, KY
* Agree to research protocol
* No allergy to either NeurOS or INOVS pads

Exclusion Criteria:

* Refusal to participate
* Emergency surgery
* Intubated and ventilated before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygenation readings from INVOS and NeurOS | From the beginning of surgery to skin closure
  Cerebral oxygenation readings from INVOS and NeurOS

SECONDARY OUTCOMES:
NeurOS brain blood volume | From the beginning of surgery to skin closure
  NeurOS brain blood volume
30 day mortality | within 30 days of surgery
  30 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jiapeng Huang, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No